CLINICAL TRIAL: NCT00005428
Title: Familial Aggregation of Stress Response
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4346; R03HL050679 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To perform data analyses on the familial aggregation of the stress response as it relates to hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Given recent advances in the analyses of genetic epidemiologic data, the database presented a unique opportunity to address timely issues pertinent to the contribution of genetic and environmental factors to individual differences in cardiovascular reactivity.

DESIGN NARRATIVE:

Secondary data analyses were performed on family data obtained in an ongoing hypertension genetic study conducted at the University of Utah with Roger R. Williams as principal investigator. The available data represented one of the largest studies of cardiovascular reactivity among genetically related individuals. During 1981-83, a total of 2,548 subjects, members of 98 extended families (multiple generations and multiple nuclear families) participated in an extensive cardiovascular examination and were assessed on a comprehensive battery of cardiovascular tests. Annual follow-up questionnaires obtained information about the onset of hypertension and new medication prescribed. In 1991-92, a follow-up exam was conducted on 1,500 subjects.

The data analysis attempted to confirm or refute hypotheses postulating a reactivity-hypertension association; investigated whether there was a sex limitation in the genetic and environmental determinants of reactivity; explored genotype-by-age interactions in the control of reactivity;and determined whether there was shared genetic and/or environmental variance between reactivity and other recognized cardiovascular risk factors such as obesity or lipids.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-08; Study Completion 1995-07 (Actual)

REFERENCES:
- [Background] Cheng LS, Carmelli D, Hunt SC, Williams RR. Segregation analysis of cardiovascular reactivity to laboratory stressors. Genet Epidemiol. 1997;14(1):35-49. doi: 10.1002/(SICI)1098-2272(1997)14:13.0.CO;2-4. PMID 9055060
- [Background] Cheng LS, Carmelli D, Hunt SC, Williams RR. Evidence for a major gene influencing 7-year increases in diastolic blood pressure with age. Am J Hum Genet. 1995 Nov;57(5):1169-77. PMID 7485169